CLINICAL TRIAL: NCT04329871
Title: An Analysis of Medtronic 670G Insulin Pump Use in Clinical Practice and the Impact on Glycemic Control, Quality of Life, and Compliance
Brief Title: Medtronic 670G Insulin Pump and the Impact on Glycemic Control, Quality of Life, and Compliance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Metabolic Research Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MetabolicRI
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analyze the Medtronic 670g pump on glycemic control

DETAILED DESCRIPTION:
An Analysis of the Medtronic 670g Insulin pump use in clinical practice and the impact on glycemic control , quality of life, and compliance

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* Documented History of Type 1 Diabetes Mellitus
* 3 months continuous use of the Medtronic 670g pump system
* given written informed consent

Exclusion Criteria:

* Less than 3 months use of the Medtronic 670g pump system
* Taking any other medication, other than the insulin used in the Medtronic 670g pump, to manage their diabetes
* having medical conditions or taking medications that would preclude subject involvement or affect the outcomes being measured, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who enter the study at Visit 1 and meet all the inclusion criteria and none of the exclusion criteria will be eligible to sign informed consent to have their data collected and analyzed
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-03-23 (Estimated); Study Completion 2021-03-23 (Estimated)

PRIMARY OUTCOMES:
Glycemic control while using the Medtronic MiniMed 670g system | through study completion, an average of 1 year.
  HbA1c, fructosamine, and glycomark will be compared between the participants last visit on previous insulin therapy and the last visit using the pump

SECONDARY OUTCOMES:
Efficacy of Quality of Life and satisfaction while using the MiniMed 670g system | through study completion, an average of 1 year
  Diabetes Treatment Satisfaction, Diabetes-dependent Quality of Life, and Pump QOL vs Previous Therapy Questionnaires will be completed by each study participant

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Horowitz, MD, Principal Investigator — Metabolic Research Institute, Inc.
Locations (1):
- Metabolic Research Institute, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
An article will be written and submitted in a major journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months to 1 year
Access Criteria: Company website
URL: http://metabolic-institute.com

REFERENCES:
- [Background] There are no Citations
- See also: Company website — http://Metabolic-institute.com
- Available data/document: Individual Participant Data Set — http://Metabolic-institute.com